CLINICAL TRIAL: NCT03242850
Title: Assuring Patient-centered Literacy Promotion for Underserved Children to Promote School Readiness
Brief Title: Assuring Patient-centered Literacy Promotion for Underserved Children Study
Acronym: APLUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Principal Investigator, Manuel E. Jimenez, MD, MS, Assistant professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro20170000878; 73308 (Other Grant/Funding Number: Robert Wood Johnson Foundation)
Record Dates: First submitted 2017-08-04; First posted 2017-08-08 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Literacy
Keywords: Reading; Text Messages; Video; Cognitive Development; Child Development; Infants
MeSH Terms: conditions — Literacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regular care group (No Intervention): This group will receive regular care including standard guidance on shared reading. Participants in this arm will not view the video at the time of enrollment nor will they receive the text messages throughout the 6 months of the randomized controlled trial.
- Intervention group (Experimental)
  Interventions: Behavioral: Intervention Group

INTERVENTIONS:
Behavioral: Intervention Group — This group will view a video on shared reading upon enrollment, receive standard guidance on shared reading, and receive a series of text messages for a period of 6 months.
  Arms: Intervention group

SUMMARY:
This study tests whether an enhanced primary cared based literacy promotion intervention consisting of a video and text message will increase shared reading occurrences between parents and children compared to the standard version.

DETAILED DESCRIPTION:
This is a randomized controlled trial aimed at assessing the effectiveness of an enhanced intervention consisting of a video and a series of text messages in promoting shared reading between parents and children. Participants will be randomized to one of two study arms (1) the enhanced intervention consisting of a video in the waiting room, standard guidance on shared reading, and a series of text messages (2) regular care which includes standard guidance on shared reading. The primary outcome will be shared reading occurrences. Secondary outcomes will include receipt of intervention, measure of the cognitive home environment, developmental screening results, and measure of parent reading beliefs.

ELIGIBILITY:
Inclusion Criteria:

1. primary caregiver of a child age 6-15 months,
2. primary language English or Spanish,
3. cell phone ownership,
4. age ≥18 years,
5. willing to receive text messages, and
6. willing to accept randomization

Exclusion Criteria:

1. Individuals unable to provide consent
2. Individuals who do not meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2019-08-24 (Actual); Study Completion 2019-08-24 (Actual)

PRIMARY OUTCOMES:
Reading Recall | Visit 2 (approx. 6 months)
  Parents will report reading occurrences in a 1 week period including a 24-hour recall.

SECONDARY OUTCOMES:
Survey of Wellbeing of Young Children Milestones | Visit 2 (approx. 6 months)
  Parents will complete the SWYC milestones, a validated, 10 item parent report, developmental screening tool.
StimQ2 Read Scale / Parental Verbal Responsivity Scale | Visit 2 (approx. 6 months)
  The StimQ2 is a parent reported measure of the cognitive home environment for children age 5 months to 6 years that assesses 4 domains: (1) Availability of Learning Materials (2) Reading (3) Parent Involvement in Developmental Advancement (4) Parental Verbal Responsiveness.
Parental Reading Beliefs Inventory | Visit 2 (approx. 6 months)
  Measure of parent reading beliefs
Receipt of intervention | Visit 2 (approx. 6 months)
  Parent report of receipt of guidance on shared reading

CONTACTS AND LOCATIONS:
Locations (1):
- Eric B. Chandler Health Center, New Brunswick, New Jersey, United States

REFERENCES:
- [Derived] Jimenez ME, Crabtree BF, Hudson SV, Mendelsohn AL, Lima D, Shelton PA, Veras J, Lin Y, Pellerano M, Morrow L, Strom BL. Enhancing Reach Out and Read With a Video and Text Messages: A Randomized Trial in a Low-Income Predominantly Latino Sample. Acad Pediatr. 2021 Aug;21(6):968-976. doi: 10.1016/j.acap.2021.02.011. Epub 2021 Feb 19. PMID 33618060